CLINICAL TRIAL: NCT00261339
Title: PRISM: Determination of the Performance Characteristics of ReQuest (TradeMark) in Practice in the Stepped Down Management of GORD
Brief Title: Determination of a Questionnaire After Treatment With Pantoprazole at Full Dose and Half Dose in Adult Patients With Symptoms of Acid Reflux (Gastroesophageal Reflux Disease) (BY1023/UK-506)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BY1023/UK-506
Record Dates: First submitted 2005-12-02; First posted 2005-12-05 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2006-12

CONDITIONS: Gastroesophageal Reflux; GERD; GORD
Keywords: Gastroesophageal Reflux; Gastroesophageal Reflux Disease; Pantoprazole
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Pantoprazole

INTERVENTIONS:
Drug: Pantoprazole

SUMMARY:
Gastroesophageal reflux disease (GERD) is a medical condition affecting the stomach and esophagus. GERD occurs when the lower esophageal sphincter does not close properly and stomach contents leaks back (refluxes) into the esophagus. GERD is one of the most common medical disorders, with estimates of up to 50% of adults reporting reflux symptoms. Proton pump inhibitors such as pantoprazole, can relieve symptoms of GERD in a large proportion of patients.

Of particular interest in GERD is the assessment of symptom severity and quality of life, and the response to treatment. Therefore, a questionnaire was developed to assess GERD symptoms ('ReQuest TradeMark in Practice'). An important point to consider when using such a questionnaire is to follow the patients´ medical response to treatment and note whether a patient needs to change dosing, such as changing from full dose to half dose, or vice versa.

The aim of the study is to determine the value of the questionnaire ('ReQuest TradeMark in Practice') according to treating physicians' clinical judgment when using pantoprazole at full and half dose. The study duration consists of a pre-treatment periods (0-2 weeks) and two treatment period (8 weeks each). During the first treatment period, pantoprazole will be administered once daily at full dose (40 mg). During the second treatment period, pantoprazole will be administered once daily at half dose (20 mg). The study will provide further data on safety and tolerability of pantoprazole.

ELIGIBILITY:
Main inclusion criteria:

* Written informed consent
* Outpatients of at least 18 years of age
* GERD
* Patients with symptoms of GERD

Main exclusion criteria:

* Signs, indicating other gastrointestinal diseases
* Other concomitant diseases
* Special restrictions for female patients
* Previous medication
* Concomitant medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2005-08

PRIMARY OUTCOMES:
GERD symptom score after 8 weeks of treatment (prior to stepping down from full dose to half dose) for patients not being symptomatically relieved from GERD after 16 weeks of treatment

SECONDARY OUTCOMES:
Symptom relief rates
symptom status (compared with pre-treatment)
time to reach first relief from reflux disease related symptoms
time to reach sustained symptom relief
relief rates from reflux disease related complaints
influence of the H. pylori-status on the symptom relief rates
safety.

CONTACTS AND LOCATIONS:
Overall Officials: Professor of Primary Care, Principal Investigator — Centre for Primary and Community Care, Sunderland, United Kingdom
Locations (41):
- United Kingdom (41):
  - Altana Pharma/Nycomed, Antrim
  - Altana Pharma/Nycomed, Ashford
  - Altana Pharma/Nycomed, Aston Clinton, Aylesbury
  - Altana Pharma/Nycomed, Atherstone, Warwick
  - Altana Pharma/Nycomed, Bangor, Northern Ireland
  - Altana Pharma/Nycomed, Barry
  - Altana Pharma/Nycomed, Barry, Vale of Glamorgan, Cardiff
  - Altana Pharma/Nycomed, Bath
  - Altana Pharma/Nycomed, Belfast
  - Altana Pharma/Nycomed, Bexhill-on-Sea, Easr Sussex
  - Altana Pharma/Nycomed, Blackpool
  - Altana Pharma/Nycomed, Bradford on Avon, Wiltshire
  - Altana Pharma/Nycomed, Cardiff (Wales)
  - Altana Pharma/Nycomed, Chesterfield
  - Altana Pharma/Nycomed, Chippenham
  - Altana Pharma/Nycomed, Chippenham, Wiltshire
  - Altana Pharma/Nycomed, Cookstown
  - Altana Pharma/Nycomed, Crawley
  - Altana Pharma/Nycomed, Crawley, West Sussex
  - Altana Pharma/Nycomed, Downpatrick, Northern Ireland
  - Altana Pharma/Nycomed, Dronfield
  - Altana Pharma/Nycomed, Ely
  - Altana Pharma/Nycomed, Glasgow
  - Altana Pharma/Nycomed, Hull
  - Altana Pharma/Nycomed, Kent
  - Altana Pharma/Nycomed, Keresely End, Coventry
  - Altana Pharma/Nycomed, Leigh Lancs
  - Altana Pharma/Nycomed, Leigh on Sea, Essex
  - Altana Pharma/Nycomed, Lisburn
  - Altana Pharma/Nycomed, Middlesex
  - Altana Pharma/Nycomed, New Street, Ledbury
  - Altana Pharma/Nycomed, Saint George's Way, Sunderland
  - Altana Pharma/Nycomed, Sheffield
  - Altana Pharma/Nycomed, Slough, Berks
  - Altana Pharma/Nycomed, Somerset
  - Altana Pharma/Nycomed, Southdown, Bath
  - Altana Pharma/Nycomed, Sunbury on Thames, Middlesex
  - Altana Pharma/Nycomed, Trowbridge
  - Altana Pharma/Nycomed, Trowbridge, Wilts
  - Altana Pharma/Nycomed, Warminster Wiltshire
  - Altana Pharma/Nycomed, Watford